CLINICAL TRIAL: NCT04230629
Title: Evaluation of Physiological Responses at the Anterior Surface of Two (Hydrophobic Acrylic) Intraocular Lens Models
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Rupert Menapace, Clinical Professor, Medical University of Vienna
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2060/2019
Record Dates: First submitted 2020-01-10; First posted 2020-01-18 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Age Related Cataracts

STUDY DESIGN:
Intervention Model Description: The investigational devices are approved intraocular lenses (IOLs) intended to be implanted after phacoemulsification in individuals suffering from age-related cataract with the need of cataract surgery. Cataract surgery with precedent bilateral IOL implantation will be performed in subjects who have signed an informed consent form. Postoperative examinations will be implemented in accordance with the approved Investigational Plan on subjects and includes: visual acuity, slitlamp examination.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vivinex XY1 (Active Comparator): Implantation of an intraocular lens Hoya Vivinex XY1
  Interventions: Device: Vivinex XY1
- Vivinex XY1A (Active Comparator): Implantation of an intraocular lens Hoya Vivinex XY1A
  Interventions: Device: Vivinex XY1A

INTERVENTIONS:
Device: Vivinex XY1 — Implantation of an intraocular lens Hoya Vivinex XY1
  Arms: Vivinex XY1
Device: Vivinex XY1A — Implantation of an intraocular lens Hoya Vivinex XY1A
  Arms: Vivinex XY1A

SUMMARY:
On the day of surgery, the the eye with astigmatism of at least 0.75dpt receives a Vivinex XY1A , HOYA Surgical Optics GmbH and the second eye to be operated receives an XY1, HOYA Surgical Optics GmbH.

A complete biomicroscopic examination and visual acuity testing using autorefractometer, will be performed 1 week (7-14days), 6 weeks (30-60days) and 5 month (4-6months) postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral age-related cataract for which phacoemulsification extraction and posterior IOL implantation is planned
* Age 40 and older
* Astigmatism of at least 0.75Diopters in one eye
* Normal findings in medical history and physical examination unless the investigator considers an abnormality to be clinically irrelevant

Exclusion Criteria:

* Diabetes mellitus
* Pseudoexfoliation syndrome
* Systemical anticoagulation
* Antiphlogistic therapy
* Antiglaucomatosa
* Uncontrolled systemic or ocular disease
* Preceding ocular surgery or trauma
* Intraoperative complications
* Pregnancy/Nursing
* Concurrently participating in any other clinical trial or if they have participated in any other clinical trial during the last 30 days

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-03-15 (Estimated); Primary Completion 2021-12-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of FBGC (foreign body giant cells) (slitlamp examination) | 5 months
  The number of foreign body giant cells on the IOLs will be assessed.

SECONDARY OUTCOMES:
Incidence of Monocytes (slitlamp examination) | 5 months
  The number of monocytes on the IOLs will be assessed. The following classification will be used: + = fewer than 10 cells/mm2; ++ = 10 to 25 cells/mm2; +++ = more than 25 cells/mm2
PCO Score (slitlamp examination) | 5 months
  Incidence and development of posterior capsular opacification will be subjectively graded: 0-10 (0= no PCO, 10= maximum PCO)
Grade of Anterior Fibrosis (slitlamp examination) | 5 months
  Grade of anterior fibrosis assessed subjectively at the slitlamp (grade 0=no fibrosis, grade 3=maximum fibrosis)
Anterior chamber reaction (slitlamp examination) | 5 months
  Incidence of cells and tyndall in the anterior chamber (ratet as - to +++ respectively)

IPD SHARING:
Plan to Share IPD: No